CLINICAL TRIAL: NCT03985917
Title: "Grupos de Canto Para Seniores" Despacho Nº 11409-C/2017, Projeto n.º 626, From Orçamento Participativo Portugal, Ministério da Cultura
Brief Title: Singing Groups for Seniors: Well-Being, Cognitive Function and Health
Acronym: Sing4Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iolanda Costa Galinha (Other)
Collaborators: DGArtes - Direção Geral das Artes (Unknown); CIS-Iscte - Centro de Investigação e Intervenção Social (Unknown)
Responsible Party: Sponsor-Investigator, Iolanda Costa Galinha, Associate Professor, Universidade Autónoma de Lisboa
Organization: Universidade Autónoma de Lisboa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Project 626 Sing Group Seniors
Record Dates: First submitted 2019-05-29; First posted 2019-06-14 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Cognitive Function; Well-Being; Physical Function; Respiratory Function; Memory; Biomarker; Anxiety; Depression; Stress; Quality of Life; Loneliness; Social Identification; Blood Pressure; Blood Glucose; Cholesterol; C-reactive Protein; Erythrocyte Sedimentation Rate; Balance; Sleep; Pain Perception; Medication Compliance; Health Complaint, Subjective; Body Weight
Keywords: Singing Group; Choir; Intervention; Older Adults; Well-Being; Cognitive Function; General Health
MeSH Terms: conditions — Respiratory Aspiration; Anxiety Disorders; Depression; Social Identification; Medication Adherence; Body Weight

STUDY DESIGN:
Intervention Model Description: Participants were recruited by invitation in the day-care centers, nursing homes and home care units run by Santa Casa da Misericórdia (a Portuguese Charity Institution, partner in the project). All older adults received an invitation with a brief description of the program and the study. In case they were interested in participating, they were invited to a meeting where the musical intervention team provided additional information about the intervention and clarified any questions from the participants. At the end of the session a detailed informed consent was signed.
Who Masked: Outcomes Assessor
Masking Description: Participants, singing group facilitators and researchers conducting the study cannot be blinded to allocation. However, the collection of the data, namely, cognitive, psychosocial, motor and physiologic outcome measures will be assessed by independent researchers, blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Singing Group Program (Experimental): Singing group intervention program that includes six components: (1) vocal warm-up exercises; (2) vocal technique; (3) rehearsal of repertoire; (4) break for socialization; (5) creation and presentation of a show; (6) assessment of participants performance (vocal tuning).
  Interventions: Other: Singing Group Intervention Program
- Alternative Social and Leisure Activities (Active Comparator): While the experimental group is participating in the intervention program, the control group will participate in the other activities proposed by the day care centers, which will be registered.
  Interventions: Other: Alternative Social and Leisure Activities

INTERVENTIONS:
Other: Singing Group Intervention Program — Each session will start with (1) relaxation, vocal warm-up and breething exercises; (2) vocal technique training; (3) memorization and interpretation of music and lyrics; (4) session breaks of 20 minutes for socialization; (5) preparation of a final choir show; (6) vocal tuning tests.
  Other Names: Choir Intervention Program
  Arms: Intervention Singing Group Program
Other: Alternative Social and Leisure Activities — Day care centers provide social and leisure activities opportunities for older adults. The control group is free to enroll in these activities.
  Other Names: Social and Leisure Activities
  Arms: Alternative Social and Leisure Activities

SUMMARY:
The researchers' implement and measure the effects of a singing group intervention program for older adults, with an RCT design, in a natural context, on the health, well-being and cognitive function of older adults.

DETAILED DESCRIPTION:
Background: Singing is a multimodal activity that requires physical, cognitive and psychosocial performance, with benefits in various domains of health and well-being of older adults. In recent years, research has increasingly studied group singing as an important cost-effective intervention to promote active and healthy aging. However, the specific factors responsible for these benefits need further experimental support, as most studies do not allow for causal inferences. This study responds to the need for further randomized controlled trials (RCT), with follow-up measurement, on the benefits of group singing in older adults with diverse socioeconomic status. Also, while most studies often focus on specific outcome measures dimensions, in this study, the conjoint effects of physical, psychosocial, emotional and cognitive dimensions are analyzed, testing mediation and moderation effects of psychosocial and cognitive variables in the health and well-being of the participants. Methods: The team implements and measures the effects of a singing group program for older adults, with an RCT design, in a natural context, before and after the intervention and in a follow-up, four months after the intervention. Participants: 140 retired older adults (> 60 years), users of a social care institution, were invited to participate in a singing group program and randomly allocated to an experimental intervention group (n = 70), and a control (n = 70) group enrolled in the regular activities proposed by the institution. The intervention consists of 34 bi-weekly group singing sessions, of two-hours each, for four months. Measures on social and emotional well-being, cognitive function, and health indicators (as blood pressure, glycemia, cholesterol, c-reactive protein, erythrocyte sedimentation rate, respiratory function, body balance, body activity, sleep quality, medication intake, and health services attendance) will be collected. Interviews on the motivation and perceived benefits of participation will also be collected. Discussion: Significant improvements are expected in the outcome measures in the experimental group after the intervention, in comparison with the control group and the pretest, validating the singing group program as a cost-effective intervention for healthy aging. Psychoemotional, psychosocial and cognitive variables are expected to be mediators of the effects of the program on the health and well-being of the participants.

ELIGIBILITY:
Inclusion criteria:

* Being 60 years old or older;
* Retired;
* Accept the invitation to participate in the singing group program;
* Not having participated in other intervention programs in the previous four months.

Exclusion criteria:

* Having a severe impairment, that is disabling for the participation in the singing group activity (e.g. severe cognitive, auditory, visual or mobility impairments).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Quality of Life - WHOQOL-BREF | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  The WHOQOL-BREF measures the subjective perception of quality of life. It consists of 26 items, of which two items measure global quality of life and 24 items measure four dimensions. In this study the (1) Physical health, (2) Psychological Health, (3) Social relationships will be measured. The items are answered in a 5 point scale, from 1 (Very Bad; Very Unsatisfied; Nothing; Never) to 5 (Very Good; Very Satisfied; Extremely; Always).
Quality of Life - WHOQOL-OLD | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  The WHOQOL-OLD measures the quality of life specifically for older adults, with 28 items, measuring six dimensions. In this study the dimensions (1) sensory abilities; (2) autonomy; (3) past, present, and future activities; and (4) social participation will be measured. The items are answered in a 5-point scale, from 1 (Nothing; Very Bad; Very Unsatisfied) to 5 (Extremely; Very Good; Very Satisfied).
Depression, Anxiety and Stress - Dass 21 | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  The DASS 21 measures Anxiety, Depression and Stress. Consists of 21 items distributed in 3 subscales of 7 items each, answered on a 4-point scale, ranging from: 0 "It did not apply to me", to 3 "Applied to me most of the time".
Positive and Negative Affect - PANAS | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  Measures the frequency of positive and negative emotions, during the past four months, and consists of two scales with 10 items each, answered on a 5-point scale from: 1 "nothing or very slightly"; to 5 "extremely".
Life Satisfaction - SWLS | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  Measures satisfaction with life in general, according to the persons' criteria. Consists of five items, answered on a 5-point scale from: 1 = strongly disagree; to 5 - I agree very much.
Self-Esteem - RSES | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  Measures the appreciation of self-worth and self-acceptance, with 10 items, answered on a 4-point Likert scale, from: 1 = strongly disagree; to 4 = strongly agree.
Loneliness - UCLA Loneliness Scale | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  Measures the feeling of being cut off from others, with four items, derived from the longer version of the ULS-20, answered on a 4-point scale from: 0 (Never), to 4 (Often / Many Times).
Social Identification - FISI | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  Measures the emotional evaluation of the relationship between the self and the ingroup, with four items, answered on a 7-point scale, ranging from: 1 "strongly disagree", to 7 "strongly agree".
Social Well-Being - Scale of Social Well-Being | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  Measures a multidimensional construct of social well-being including the dimensions: social acceptance, social coherence, social actualization, social integration and social contribution. Constituted by 33 items, answered on a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree).
Cognitive Function - MoCA | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  Measures six cognitive functions: executive function; visuospatial skills; short-term memory; language; attention, concentration and working memory; and temporal and spatial orientation. The test is constituted by six groups of tasks and exercises. The maximum score is 30 points; higher scores indicate better cognitive performance.
Short-term auditory verbal memory - RAVELT | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  The scale measures the rate of verbal learning, learning strategies, retroactive, and proactive interference, presence of confabulation or confusion in memory processes, retention of information, and differences between learning and retrieval. It consists of a list of 15 unrelated words repeated over five different trials, which participants are asked to repeat.
Attention and Executive Function - Trail Making Test | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  The test measures the processing speed, mental flexibility, and divided attention. It consists of a task of connecting a trail of numbers with a drawing line. In this study, TMT A will be used, providing two direct scores: time to complete part A and performance errors.
Processing Speed - Digit Symbol Test | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  The test measures the processing speed of non-verbal information. It consists of a task of drawing figures corresponding to numbers. It also measures cognitive and motor speed, planning ability, visual memory, visuomotor coordination, motivation to perform the task and attention.
Blood Pressure - Licensed laboratory | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  Measures the pressure with which the blood circulates within the arteries. Data collected and analyzed by a licensed laboratory.
Pulse - Licensed laboratory | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  The count of arterial pulse per minute, measures the number of times the heart beats per minute. Data collected and analyzed by a licensed laboratory.
Glycemia - Blood sample - Licensed laboratory | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  Measures the amount of glucose present in the blood, used in the diagnosis and treatment of several diseases as diabetes mellitus or hypoglycemia. Data is collected and analyzed by a licensed laboratory.
Cholesterol - Blood sample - Licensed laboratory | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  Measures total cholesterol, a fatty substance produced by the liver, present in all body cells and essential for the formation of the cell membranes hormone synthesis, digestion of fats, production of bile, metabolism of vitamins A, D, E and K, important in the constitution of global coronary disease risk. Data is collected and analyzed by a licensed laboratory.
C-reactive protein (CRP) - Blood sample - Licensed laboratory | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  Measures C-reactive protein, a protein produced in the liver and in case of inflammatory states its production increases. Indicates an ongoing, but not specific, organism infection. It can also be high in case of neoplasia. Data collected and analyzed by a licensed laboratory.
Erythrocyte Sedimentation Rate (ESR) - Blood sample - Licensed laboratory | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  A measure of the red blood cells sedimentation by micro photometry over a period of time. A blood sedimentation rate is tested to detect inflammation in the body or to follow the progress of a disease. Data is collected and analyzed by a licensed laboratory.
Body Weight - Professional scale | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  Body weight is assessed by weighing the person with light clothing, without shoes and while fasting.
Respiratory Function - Spirometry (Medikro Pro) - Air Volume | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  The test consists of a simple examination, which allows to globally evaluate how the lungs are functioning by measuring the volume of air (measured in litres with the tests FVC, FEV1 and FEV6). In addition the Tiffeneau-Pinelli Index will be measured, which is a ratio between FVC and FEV1. Data is collected by trained researchers in motricity sciences.
Respiratory Function - Spirometry (Medikro Pro) - Air Speed | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  The test consists of a simple examination, which allows to globally evaluate how the lungs are functioning by measuring the speed of air expired (litres per second, measured with the tests PEF, FEF 25 to 75%). Data is collected by trained researchers in motricity sciences.
Body Balance - Unipedal Stance Test. | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  The participant is instructed to balance on a foot of their choosing for up to 20 seconds. The number of seconds in balance is registered as the score of this test. Data collected by trained researchers in motricity sciences.
Physical Activity - Actigraphy (GT3X accelerometer) | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  Actigraphy registers the body accelerations in three axes (vertical, antero-posterior, and medio-lateral). Participants will be asked to wear the accelerometer around the hip for seven consecutive days (day and night, except when bathing). The accelerometer provides a measure of the frequency, intensity, and duration of physical activity and allows for the classification of activity levels as sedentary, light, moderate and vigorous.
Sleep Quality - Actigraphy (GT3X accelerometer) | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  Actigraphy registers the body accelerations in three axes (vertical, antero-posterior, and medio-lateral). Participants will be asked to wear the accelerometer around the hip for seven consecutive days (day and night, except for bathing). The accelerometer provides a measure of the frequency, intensity, and duration of physical activity and allows for a measure of the total duration of sleep.
Pain Perception - The Brief Pain Inventory, | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  The scale measures different types of pain, with nine questions: a first one that is optional; a second one based on drawings of the human body to locate the pain in the body; four items about pain intensity (worst pain, least pain, average pain, pain right now); two items on pain relief or medication; and one item on pain interference, with seven sub-items (general activity, mood, walking ability, normal walk, relations with other people, sleep, and enjoyment of life). Answering options from: 0 "No pain / Did not interfered"; and 10 "The greatest pain possible / Completely interfered".
Medication Intake - Social Support Institution | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  Medication and dosage are registered and supplied by the Social Care Institution to the research team with the authorization of the participants.
Health Services Attendance - Social Support Institution | Change from baseline at 4 months (post-test) and at 10 months (follow-up).
  Number and type of health services appointments registered and supplied by the Social Care Institution to the research team with the authorization of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Iolanda C. Galinha, Ph.D,, Study Director — Universidade Autónoma de Lisboa
Locations (1):
- Universidade Autónoma de Lisboa, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Galinha IC, Garcia-Martin MA, Lima ML. Sing4Health: Randomised controlled trial of the effects of a singing group program on the subjective and social well-being of older adults. Appl Psychol Health Well Being. 2022 Feb;14(1):176-195. doi: 10.1111/aphw.12297. Epub 2021 Aug 10. PMID 34378330
- [Derived] Galinha IC, Fernandes HM, Lima ML, Palmeira AL. Intervention and mediation effects of a community-based singing group on older adults' perceived physical and mental health: the Sing4Health randomized controlled trial. Psychol Health. 2023 Jan;38(1):73-93. doi: 10.1080/08870446.2021.1955117. Epub 2021 Aug 6. PMID 34355628
- [Derived] Galinha IC, Farinha M, Lima ML, Palmeira AL. Sing4Health: protocol of a randomized controlled trial of the effects of a singing group intervention on the well-being, cognitive function and health of older adults. BMC Geriatr. 2020 Sep 18;20(1):354. doi: 10.1186/s12877-020-01686-6. PMID 32948120
- See also: Projeto n.º 626, from Orçamento Participativo Portugal, Ministério da Cultura — https://dre.pt/home/-/dre/114422404/details/maximized